CLINICAL TRIAL: NCT01955993
Title: The Pharmacokinetics of Intravenous Fentanyl in Adolescent Patients With Higher BMI Percentiles.
Brief Title: Fentanyl Metabolism in Obese Adolescents
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Janelle Vaughns, Assistant Professor, Anesthesiology and Perioperative Medicine, Children's National Research Institute
Other Study IDs: 1809
Record Dates: First submitted 2013-09-23; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Morbid Obesity
Keywords: Obesity, adolescence,pharmacokinetics,fentanyl
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fentanyl use for surgical pain: Adolescent patient having surgery

SUMMARY:
Fentanyl is a frequently used pain medication in pediatric and adult anesthesia. Although there are some studies considering the breakdown of oral, transmucosal and intravenous fentanyl preparations in children, the disposition of fentanyl in pediatric patients has not been sufficiently described. This study aims to show that the clearance of fentanyl in obese children and adolescents is increased as compared to children with a normal weight. Consequently, the elimination half-life of fentanyl is different in overweight and obese children from that in children having a normal body weight.

DETAILED DESCRIPTION:
Obesity represents one of the most important public health issues according to the World Health Organization. It has reached epidemic proportions globally, with approximately 1.5 billion overweight adults 20 years and older and at least 600 million of them clinically obese in 2008. According to the most recent NHANES survey (2003-2006), over two-third of the adults in the US are overweight or obese (overweight 68%, half of them obese) and about 17.6% of children and adolescents aged 12 to 19 were considered overweight or obese.

Obesity has also become an important challenge for the anesthesiologist. Safety and drug dosing particularly within the field of pediatric anesthesia, is of paramount concern as it can affect patient outcomes. Data collected in the United Kingdom from more than 100,000 anesthetized pediatric patients showed that a critical incident is twice as likely to occur in an obese child in the preoperative period as in an obese adult. A possible explanation may be linked to the lack of precision in drug dosing for these obese patients.

Fentanyl is a frequently used opioid analgesic in pediatric and adult anesthesia. Fentanyl is commonly administered to pediatric patients undergoing anesthesia as it is has a high potency, a rapid onset and a short duration of action. Due to these properties intravenously administered fentanyl is well suited as an analgesic compound in general anesthesia in pediatric patients.

The pharmacokinetics of fentanyl in adults have been well documented. Although there are some studies investigating the pharmacokinetic properties of oral, transmucosal and intravenous fentanyl preparations in children, the disposition of fentanyl in pediatric patients has not been sufficiently described. Several studies in infants and children report age-dependent differences in the pharmacokinetic/ pharmacodynamic parameters of intravenously administered fentanyl.

Currently there are no data available about the pharmacokinetics/ pharmacodynamics of fentanyl in adolescent obese patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject will be an inpatient or outpatient admitted for at least 24 hours observation as part of the surgical plan of care

  2. The BMI will be calculated using height and weight and will include the 5th to 84th percentile for the control group and greater than or equal to 95th percentile for the obese adolescents.

  3. All racial and ethnic groups will be included.

Exclusion Criteria:

1. Any patient that is pregnant or lactating.
2. Prior exposure to any opioid including fentanyl within a 24 hour period.
3. Patients with known hypersensitivity to any opioids.
4. History of central nervous system dysfunction and active upper airway disease and liver and renal disease. Patients diagnosed with renal or liver disease as evidenced by abnormal function tests within the past 12 months will be excluded.
5. Patients who are treated with drugs known to affect the cytochrome P450 3A (CYP3A4), like antiepileptics, imidazole derivates, macrolides, corticosteroids and grapefruit juice

   -

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Single, hospital based surgical center
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Systemic clearance of fentanyl and its metabolites norfentanyl, hydroxynorfentanyl and despropionylfentanyl in adolescent surgical patients with higher BMI percentiles. | two years

SECONDARY OUTCOMES:
to determine the frequency of the CYP3A5 genotype (*1 and *3 alleles) of all participants | two years

CONTACTS AND LOCATIONS:
Overall Officials: John van den Anker, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Vaughns JD, Ziesenitz VC, Williams EF, Mushtaq A, Bachmann R, Skopp G, Weiss J, Mikus G, van den Anker JN. Use of Fentanyl in Adolescents with Clinically Severe Obesity Undergoing Bariatric Surgery: A Pilot Study. Paediatr Drugs. 2017 Jun;19(3):251-257. doi: 10.1007/s40272-017-0216-6. PMID 28238111